CLINICAL TRIAL: NCT05665335
Title: A Post-Market Study of a Minimally Invasive Beast Lift Procedure Utilizing the Renuvion APR System
Brief Title: A Post-Market Study in Greece of a Minimally Invasive Breast Lift Procedure Utilizing the Renuvion APR System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Apyx Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX-22-03-GR
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Results first posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Breast Ptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Renuvion APR System (Experimental): Subjects treated with the Renuvion APR system in both breasts.
  Interventions: Device: Renuvion APR System

INTERVENTIONS:
Device: Renuvion APR System — The treatment area is defined as superior most not to exceed a horizontal line from the superior aspect of the axilla to the midline; inferior most not to cross the junction of the breast with the abdomen (inframammary fold). Lateral border to the outermost curvature of the breast or a vertical line drawn from the preaxillary line to the IMF; medial most to the innermost curvature of the breast up to 1 cm lateral to the sternal midline. The procedure will be in the intradermal and subdermal planes in the full breast area, without penetrating the breast gland.
  Renuvion APR System settings will be 60-70% Power, 1.5 LPM, and up to 6 retrograde or 3 antegrade/retrograde passes, with a minimum of 2 incision sites.

SUMMARY:
This is a prospective, non-randomized, single-center, evaluator blinded study of up to 15 subjects undergoing a minimally invasive breast lift procedure utilizing the Renuvion APR System. Subjects will receive treatment with the Renuvion APR System to both breasts.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, single-center, evaluator blinded study of up to 15 subjects undergoing a minimally invasive breast lift procedure utilizing the Renuvion APR System. Subjects will receive treatment with the Renuvion APR System to both breasts.

At baseline, the grade of breast ptosis, breast measurements and pre-surgery photographs will be taken using the site's camera system.

Procedure data and adverse events will be captured.

Follow-up visits will occur at 30, 90, and 180-days post-procedure. Subjects may also be seen back for follow-up at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects, ages 18 - 75 years old.
* ASA Physical Status Classification System Class I and Class II subjects.
* Breast Ptosis Class II and Class III as per the Eyck et al, Rainbow Scale for Assessing Breast Ptosis.
* Breast Cup Size A and Size B.
* Understands and accepts the obligation not to undergo any other procedures or treatments in the areas to be treated during study participation.
* Absence of physical conditions unacceptable to the investigator.
* Females of childbearing potential who are sexually active must be willing to use an approved method of birth control during study participation.
* Willing and able to comply with protocol requirements, including study-required images/photos, assessments/measurements, and returning for follow-up visits.
* Willing to release rights for the use of study photos, including in publication.
* Able to read, understand, sign, and date the informed consent.
* Able to communicate with the site via video and/or photographs, in the event of a virtual follow-up visit.

Exclusion Criteria:

* Subjects presenting with ASA Physical Status Classification System Classes III or higher.
* Breast ptosis Class IV or more as per the Eyck et al, Rainbow Scale for Assessing Breast Ptosis.
* Breast Cup Size C, Size D or larger.
* Prior surgery or procedure in the breast area (i.e., implants, skin tightening procedures, breast reduction, etc.).
* Pregnant, lactating, or plans to become pregnant during study participation.
* Known hypersensitivity or allergy to tumescent anesthetic (lidocaine/ epinephrine).
* Known hypersensitivity or allergy to ibuprofen or other NSAIDS.
* Previous treatment in the study treatment area.
* Active systemic or local skin disease that may alter wound healing.
* Significant or uncontrolled medical condition that in the opinion of the investigator participation in the study may compromise the patient's health.
* History of autoimmune disease (excluding Hashimoto's thyroiditis).
* Known susceptibility to keloid formation or hypertrophic scarring.
* Cancerous or pre-cancerous lesions in the area to be treated.
* Possesses a surgically implanted electronic device (i.e., pacemaker).
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Participation in any other investigational study within 30 days prior to consent and throughout study participation.
* Subject who, in the opinion of the investigator, is not an appropriate candidate for the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female subjects
Enrollment: 15 (Actual)
Dates: Start 2022-11-28 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aris Sterodimas, MD, MSc, PhD, Principal Investigator — Metropolitan General Hospital
Locations (1):
- Metropolitan General Hospital, Athens, Greece

REFERENCES:
- [Result] Sterodimas A, Moutafis A, Nicaretta B, Champsas G. A Prospective Study on Helium-Based Plasma Radiofrequency for Minimally Invasive Breast Lift Scarless Mastopexy. Aesthet Surg J Open Forum. 2025 Mar 5;7:ojaf004. doi: 10.1093/asjof/ojaf004. eCollection 2025. PMID 40236884

RESULTS

PARTICIPANT FLOW:
Groups:
- Renuvion APR System: Subjects treated with the Renuvion APR system in both breasts.
  Renuvion APR System: The treatment area is defined as superior most not to exceed a horizontal line from the superior aspect of the axilla to the midline; inferior most not to cross the junction of the breast with the abdomen (inframammary fold). Lateral border to the outermost curvature of the breast or a vertical line drawn from the preaxillary line to the IMF; medial most to the innermost curvature of the breast up to 1 cm lateral to the sternal midline. The procedure will be in the intradermal and subdermal planes in the full breast area, without penetrating the breast gland.
  Renuvion APR System settings will be 60-70% Power, 1.5 LPM, and up to 6 retrograde or 3 antegrade/retrograde passes, with a minimum of 2 incision sites.
Period: Overall Study
Arm/Group | Renuvion APR System
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Nationality: Greek | 12
  Nationality: Albanian | 1
  Nationality: Brazilian | 2
Region of Enrollment [Number; unit: participants]
  Greece | 15
Breast Cup Size [Count of Participants; unit: Participants] — Hemicircumference measured across the maximum projection of the breast from the medial inflection point to the lateral inflection point where the breast creates a crease in the skin when the breast is displaced or pushed medially or laterally. A Cup = 17.0 cm. B Cup = 19.5 cm. C Cup = 21.5 cm. D Cup = 23.5 cm. DD Cup = 25.0 cm.
  Participants
    Cup Size A | 2
    Cup Size B | 13
ASA Status [Count of Participants; unit: Participants] — Evaluation by the investigator determining patient health by the American Society of Anesthesiologists Scale:
  ASA I = A normal healthy patient ASA II = A patient with mild systemic disease ASA III = A patient with severe systemic disease ASA IV = A patient with severe systemic disease that is a constant threat to life ASA V = A moribund patient who is not expected to survive without the operation ASA VI = A declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    ASA I | 13
    ASA II | 2
Rainbow Scale for Breast Ptosis [Count of Participants; unit: Participants] — Evaluation by the investigator grading the amount of visual breast ptosis (breast laxity) by the Rainbow scale of ptosis includes 5 grades: a Grade I (no ptosis), Grade II (minimal ptosis), Grade III (moderate ptosis), Grade IV (more than moderate ptosis), V (severe ptosis) scale.
  Participants
    Grade I | 0
    Grade II | 15
    Grade III | 0
    Grade IV | 0
    Grade V | 0
Breast-Q Survey [Mean (Standard Deviation); unit: Average units on a scale] — Subjects will complete the Psychosocial Well-Being and Sexual Well-Being questionnaires. Subjects were instructed "With your breasts in mind, in the past week, how often have you felt:". Responses were 5 options: 1 - None of the time, 2 - A little of the time, 3 - Some of the time, 4 - Most of the time, 5 - All of the time.
  Average units on a scale
    Confident in a social setting? | 3.4 (0.9)
    Good about yourself? | 3.6 (0.7)
    Confident in your clothes? | 3.1 (0.6)
    Of equal worth to other women? | 3.2 (0.9)
    Attractive? | 3.2 (0.7)
    Accepting of your body? | 3.2 (0.8)
    Self-assured? | 3.7 (0.6)
    Confident about your body? | 3.0 (0.5)
    Self-confident? | 3.9 (0.4)
    Sexually attractive in your clothes? | 3.1 (0.7)
    Comfortable/at ease during sexual activity? | 3.4 (0.8)
    Confident sexually? | 3.2 (0.7)
    Sexy when unclothed? | 2.5 (0.6)
    Confident sexually about how your breasts look when unclothed? | 2.3 (0.5)
Average Reported Pain by Subject [Count of Participants; unit: Participants] — Study subjects will be asked to complete a 11-point Numeric Rating Scale (NRS) for the level of pain and discomfort associated with the study procedure. Rating Scale where 0 is "No Pain" and 10 is "Worst Possible Pain".
  Participants
    0 | 15
    1 | 0
    2 | 0
    3 | 0
    4 | 0
    5 | 0
    6 | 0
    7 | 0
    8 | 0
    9 | 0
    10 | 0

OUTCOME MEASURES:

1. Primary Outcome: Independent Photographic Review of Before and After Images Compared to Baseline Compared to D180.
Description: Improvement in breast ptosis as determined by a masked, qualitative assessment of photographs at 180-days post-treatment compared to baseline by blinded independent reviewers.
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants | 11

2. Secondary Outcome: Independent Photographic Review of Before and After Images Compared to Baseline at D90.
Description: Improvement in breast ptosis as determined by a masked, qualitative assessment of photographs at 90-days post-treatment compared to baseline by blinded independent reviewers.
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants | 10

3. Other Pre Specified Outcome: Change in Morphometric Breast Measurements at Day 30
Description: Bilateral analysis of change to Morphometric breast measurements as per Brown, An Analysis of Ptosis at baseline and at D30.
Time Frame: 30-Day
Measure: Mean (Standard Deviation); unit: cm change from baseline
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
cm change from baseline
  SNN-N: Suprasternal notch to nipple distance | -0.7 (0.5)
  IMC-N: Inframammary crease to nipple distance | -0.3 (0.5)
  MCL-N: Midclavicular line to nipple distance | -0.7 (0.5)
  NAC: nipple-areola complex diameter | -0.1 (0.4)
  PROJ: maximum point of breast projection measured perpendicular to the chest wall | -0.2 (1.2)
  N-N: nipple to nipple distance | -0.3 (1.0)
  SSN-IMC: vertical distance from the suprasternal notch to the inframammary crease | -0.5 (0.6)
  SSN-base: vertical distance from the suprasternal notch to the lowest point on the base | -0.9 (0.8)

4. Other Pre Specified Outcome: Change in Morphometric Breast Measurements at Day 90
Description: Bilateral analysis of change to Morphometric breast measurements as per Brown, An Analysis of Ptosis at baseline and at D90.
Time Frame: 90-Day
Measure: Mean (Standard Deviation); unit: cm change from baseline
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
cm change from baseline
  SNN-N: measurements taken at the mid nipple diameter on both sides | -0.9 (0.5)
  IMC-N: measurement taken from the base of the breast to the base of the nipple | -0.6 (0.6)
  MCL-N: measurement taken from the mid clavicle to the mid nipple | -0.8 (0.6)
  NAC: nipple-areola complex diameter | -01. (0.5)
  PROJ: maximum point of breast projection measured perpendicular to the chest wall | 0 (1.2)
  N-N: measurements taken at the mid nipple diameter on both sides | -0.3 (1.1)
  SSN-IMC: vertical distance from the suprasternal notch to the inframammary crease | -0.7 (0.8)
  SSN-base: vertical distance from the suprasternal notch to the lowest point on the base | -1.1 (0.8)

5. Other Pre Specified Outcome: Change in Morphometric Breast Measurements at Day 180
Description: Bilateral analysis of change to Morphometric breast measurements as per Brown, An Analysis of Ptosis at baseline and at D180.
Time Frame: 180-Day
Measure: Mean (Standard Deviation); unit: cm change from baseline
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
cm change from baseline
  SNN-N: measurements taken at the mid nipple diameter on both sides | -1.2 (0.7)
  IMC-N: measurement taken from the base of the breast to the base of the nipple | -0.6 (0.5)
  MCL-N: measurement taken from the mid clavicle to the mid nipple | -0.9 (0.7)
  NAC: nipple-areola complex diameter | 0.1 (0.4)
  PROJ: maximum point of breast projection measured perpendicular to the chest wall | 0.3 (1.2)
  N-N: measurements taken at the mid nipple diameter on both sides | 0 (1.1)
  SSN-IMC: vertical distance from the suprasternal notch to the inframammary crease | -0.8 (1.0)
  SSN-base: vertical distance from the suprasternal notch to the lowest point on the base | -1.5 (1.0)

6. Other Pre Specified Outcome: Change in Breast Ptosis Classification at Day 180
Description: Evaluation by the investigator grading the amount of visual breast ptosis (breast laxity) by the Rainbow scale of ptosis includes 5 grades: a Grade I (no ptosis), Grade II (minimal ptosis), Grade III (moderate ptosis), Grade IV (more than moderate ptosis), V (severe ptosis) scale.
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Grade I | 6
  Grade II | 9
  Grade III | 0
  Grade IV | 0
  Grade V | 0

7. Other Pre Specified Outcome: Investigator Global Aesthetic Improvement Scale (GAIS) at Day 30
Description: The investigator will grade the overall improvement of treatment area as very much improved, much improved, improved, no change, worse, much worse, or very much worse.
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 1
  Much Improved | 10
  Improved | 4
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

8. Other Pre Specified Outcome: Investigator Global Aesthetic Improvement Scale (GAIS) at Day 90
Description: as for outcome 7
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 4
  Much Improved | 9
  Improved | 2
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

9. Other Pre Specified Outcome: Investigator Global Aesthetic Improvement Scale (GAIS) at Day 180
Description: as for outcome 7
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 10
  Much Improved | 5
  Improved | 0
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

10. Other Pre Specified Outcome: Subject Global Aesthetic Improvement Scale (GAIS) at Day 30
Description: The Subject will grade overall improvement of treatment area as very much improved, much improved, improved, no change, worse, much worse, or very much worse.
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 1
  Much Improved | 11
  Improved | 3
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

11. Other Pre Specified Outcome: Subject Global Aesthetic Improvement Scale (GAIS) at Day 90
Description: as for outcome 10
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 4
  Much Improved | 8
  Improved | 3
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

12. Other Pre Specified Outcome: Subject Global Aesthetic Improvement Scale (GAIS) at Day 180
Description: as for outcome 10
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  Very Much Improved | 10
  Much Improved | 5
  Improved | 0
  No Change | 0
  Worse | 0
  Much Worse | 0
  Very Much Worse | 0

13. Other Pre Specified Outcome: Patient Satisfaction Questionnaire (PSQ) at Day 180
Description: Subjects will be asked to complete a satisfaction survey referring to the assessment of baseline photos, current photos, and a mirror. Yes/No - Did you notice any improvement in the laxity or sagginess of your breasts? If yes, checkbox - Less sagging, Breasts look higher on the chest, Nipple placement is improved, Breasts appear more youthful, and/or Other. How would you characterize your satisfaction with the treatment? - very satisfied, satisfied, slightly satisfied, neither satisfied or dissatisfied, slightly dissatisfied, dissatisfied, very dissatisfied. Yes/No - Would you recommend this treatment to your friends and family members?
Time Frame: 180-Day
Measure: Number; unit: participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
participants
  Yes, Improvement Noticed in Breast Area | 15
  Yes, Less Sagging Breasts | 15
  Yes, Breasts Look Higher on Chest | 15
  Yes, Nipple Placement is Improved | 15
  Yes, Breasts Appear More Youthful | 15
  Yes, Would recommend to friends and family | 15

14. Other Pre Specified Outcome: Breast-Q Survey
Description: Subjects will complete the Psychosocial Well-Being and Sexual Well-Being questionnaires. Subjects were instructed "With your breasts in mind, in the past week, how often have you felt:". Responses were 5 options: 1 - None of the time, 2 - A little of the time, 3 - Some of the time, 4 - Most of the time, 5 - All of the time.
Time Frame: 180-Day
Measure: Mean (Standard Deviation); unit: average units on a scale
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
average units on a scale
  Confident in a social setting? | 4.3 (0.5)
  Good about yourself? | 4.5 (0.5)
  Confident in your clothes? | 4.5 (0.5)
  Of equal worth to other women? | 4.3 (0.5)
  Attractive? | 4.2 (0.6)
  Accepting of your body? | 4.4 (0.6)
  Self-assured? | 4.4 (0.5)
  Confident about your body? | 4.5 (0.5)
  Self-confident? | 4.7 (0.5)
  Sexually attractive in your clothes? | 4.2 (0.6)
  Comfortable/at ease during sexual activity? | 4.3 (0.6)
  Confident sexually? | 4.3 (0.5)
  Sexy when unclothed? | 4.4 (0.6)
  Confident sexually about how your breasts look when unclothed? | 4.2 (0.6)

15. Other Pre Specified Outcome: Average Reported by Subject at Procedure
Description: Study subjects will be asked to complete a 11-point Numeric Rating Scale (NRS) for the level of pain and discomfort associated with the study procedure. Rating Scale where 0 is "No Pain" and 10 is "Worst Possible Pain"
Time Frame: Procedure Day 0 (within 60 minutes following treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

16. Other Pre Specified Outcome: Average Reported Pain by Subject at Day 30
Description: as for outcome 15
Time Frame: 30-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

17. Other Pre Specified Outcome: Average Reported Pain by Subject at Day 90
Description: as for outcome 15
Time Frame: 90-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

18. Other Pre Specified Outcome: Average Reported Pain by Subject at Day 180
Description: as for outcome 15
Time Frame: 180-Day
Measure: Count of Participants; unit: Participants
Arm/Group | Renuvion APR System
Number analyzed (Participants) | 15
Participants
  0 | 15
  1 | 0
  2 | 0
  3 | 0
  4 | 0
  5 | 0
  6 | 0
  7 | 0
  8 | 0
  9 | 0
  10 | 0

ADVERSE EVENTS:
Time Frame: Adverse events and expected treatment effects were evaluated over the 180-day follow-up period.
Description: Adverse events and expected treatment effects (ETEs) were collected.
Arm/Group | Renuvion APR System
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT05665335/Prot_SAP_000.pdf